CLINICAL TRIAL: NCT06612229
Title: Improvement of Methodological Approaches to Diagnostics and Tactics of Treatment of Biliary Fistulas in Surgery of Liver Echinococcosis
Brief Title: Biliary Fistulas in Surgery of Liver Echinococcosis
Acronym: BFISOLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Republican Specialized Scientific and Practical Medical Center of Surgery Named After V. Vakhidov (Other)
Responsible Party: Principal Investigator, Azam Babadjanov, Professor, Republican Specialized Scientific and Practical Medical Center of Surgery Named After V. Vakhidov
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 27022024
Record Dates: First submitted 2024-02-27; First posted 2024-09-25 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-09

CONDITIONS: Echinococcosis, Hepatic; Biliary Fistula
Keywords: Echinococcosis of the liver; Biliary fistula; Conservative surgical treatment
MeSH Terms: conditions — Echinococcosis, Hepatic; Biliary Fistula

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- operation for liver echinococcosis complicated by a biliary fistula (Other)
  Interventions: Procedure: Conservative surgical treatment of liver echinococcosis, verification of occult biliary fistulas and their elimination by weaving and using medical cyanoacrylate glue

INTERVENTIONS:
Procedure: Conservative surgical treatment of liver echinococcosis, verification of occult biliary fistulas and their elimination by weaving and using medical cyanoacrylate glue — In conservative surgical operations for liver echinococcosis, the biliary fistula is identified, onto which a U-shaped suture is applied, after which medical cyanoacrylate glue is applied between the suture stitches to the fibrous capsule in the fistula area and the suture threads are tied.

SUMMARY:
The objective of the study is to improving the results of surgical treatment of liver echinococcosis complicated by biliary fistula by optimizing diagnostic approaches to early verification of this complication and improving the tactical and technical aspects of its elimination.

ELIGIBILITY:
Inclusion Criteria:

* Age under 18 years;
* Informed consent for inclusion in the study;
* The presence of liver echinococcosis, for which conservative surgical treatment will be performed;
* The presence of the entire spectrum of necessary preoperative diagnostic measures;
* A full description of all stages of surgical intervention, indicating the type of intervention (open or laparoscopic surgery, location and size of the echinococcal cyst in the liver, type of antiparasitic treatment, presence or absence of a biliary fistula in the residual cavity, actions taken in relation to the fistula, the option of eliminating the residual cavity and drainage;
* Availability of objective data on the characteristics of the postoperative course, including dynamic indicators of the patient's condition, temperature, amount and nature of discharge through the drainage, the time of drainage removal, the type of complications (if any) and the method of their treatment, the duration of the hospital period, data on the characteristics of the posthospital period up to 3 months of observation;
* Absence of concomitant pathology that may affect the outcome of the surgery.

Exclusion Criteria:

* Age under 18 years;
* Refusal to participate in the study;
* Extrahepatic echinococcosis without liver damage;
* Absence of the full range of preoperative diagnostic data;
* Difficulties with objective analysis of the features of the performed surgical treatment;
* Incomplete data on monitoring the postoperative hospital and remote (up to 3 months) period;
* The presence of concomitant pathology that may affect the outcome of the operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-22 (Actual); Primary Completion 2026-09-22 (Estimated); Study Completion 2026-12-23 (Estimated)

PRIMARY OUTCOMES:
Measuring the incidence of bile leakage after conservative surgical interventions for liver echinococcosis | 3 months
  assessing the effectiveness of the method for eliminating biliary fistulas in the fibrous capsule during organ-preserving surgeries for liver echinococcosis, characterized by creating a two-level strengthening of the fistula area by applying U-shaped sutures and a cyanoacrylate adhesive composition
Measuring the time of closure of biliary fistulas in the postoperative period | 3 months
  In the group of patients with the development of biliary fistulas after surgery, the time of their closure in days will be studied

SECONDARY OUTCOMES:
Measuring the costs of treating patients with liver echinococcosis | 3 months
  Economic costs will be assessed for patients with liver echinococcosis who undergo conservative surgical interventions, taking into account the absence or development of bile leakage in the postoperative period
Measurement of the quality of life of patients after conservative surgical interventions for liver echinococcosis. | 3 months
  The quality of life will be analyzed using the SF-36 (The 36-Item Short Form Survey) questionnaire in patients after conservative surgical interventions, taking into account the absence or development of bile leakage in the postoperative period. It stems from a study called the Medical Outcomes Study for the objective measure of the quality of life. Scores for the various domains are transformed and combined using a scoring key to obtain a total score indicating a range from low to high quality of life (from 0 to 100 points). Scores for two components, the physical component and the mental component, can also be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Republican specialized scientific and practical medical center of surgery named after academician V.Vakhidov, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: Undecided